CLINICAL TRIAL: NCT01099657
Title: Virtual Reality Hypnosis for Chronic Pain Reduction
Acronym: VRHChP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Shelley A. Wiechman, Associate Professor, Rehabilitative Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31498
Record Dates: First submitted 2010-04-01; First posted 2010-04-07 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality Hypnosis (Experimental): Virtual Reality Hypnosis for chronic pain
  Interventions: Behavioral: Virtual Reality Hypnosis for chronic pain
- Virtual Reality Distraction (Experimental): Virtual Reality Distraction for Chronic Pain
  Interventions: Behavioral: Virtual Reality Distraction for Chronic Pain

INTERVENTIONS:
Behavioral: Virtual Reality Hypnosis for chronic pain — At the time of their clinic visit,the subject will answer pain and anxiety questionnaires before experiencing Virtual Reality Hypnosis. After VRH, the will again answer Pain and anxiety questionnaires.
  Arms: Virtual Reality Hypnosis
Behavioral: Virtual Reality Distraction for Chronic Pain — At the time of their clinic visit,the subject will answer pain and anxiety questionnaires before experiencing Virtual Reality Distraction. After VRD, the will again answer Pain and anxiety questionnaires.
  Arms: Virtual Reality Distraction

SUMMARY:
We would like to determine how well hypnosis works when induced through virtual reality medium for patients who have suffered a major burn injury in the past two years and suffer from chronic pain. These patients are coming back to the outpatient burn and plastic clinic at Harborview Medical Center for routine follow-up. We think that patients will find VR-Hypnosis interesting, and it will help them relax and feel less pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 75 years
* Able to complete subjective evaluations of pain
* English-speaking
* Able to communicate orally

Exclusion Criteria:

* Age less than 13 years or greater than 75 years
* Incapable of indicating subjective evaluation of pain
* Non-English-speaking (Virtual Reality Hypnosis only available in English)
* Demonstrating delirium, psychosis, or Organic Brain Disorder
* Unable to communicate verbally
* Significant developmental disability
* Extreme susceptibility to motion sickness
* Significant head/or neck injury
* Pregnant women

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pain and anxiety | pre and post VR and then up to one month
  The subjects will answer questions regarding pain and anxiety at the time of their clinic visit, before and after experiencing virtual reality. Then the subject will be followed for up to one month.

CONTACTS AND LOCATIONS:
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided